CLINICAL TRIAL: NCT04389645
Title: Interferon Gamma Induced Protein 10 (IP-10) in a Clinical Decision Support Protocol in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MM-5000-BV
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IP-10 in CDS protocol — Dynamic IP-10 measurements in hospitalized COVID-19 positive patients

SUMMARY:
The proposed project will pilot incorporation of rapid serial measurements of IP-10 into a CDS tool for moderate and severe COVID-19 patients.

The tool was applied to all comers with confirmed COVID-19 diagnosis at a secondary medical center in Israel.

ELIGIBILITY:
Inclusion Criteria:

* PCR- positive for COVID-19

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PCR-positive COVID-19 all comers
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
IP-10 levels | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Lev, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Lev S, Gottesman T, Sahaf Levin G, Lederfein D, Berkov E, Diker D, Zaidman A, Nutman A, Ilan Ber T, Angel A, Kellerman L, Barash E, Navon R, Boico O, Israeli Y, Rosenberg M, Gelman A, Kalfon R, Simon E, Avni N, Hainrichson M, Zarchin O, Gottlieb TM, Oved K, Eden E, Tadmor B. Observational cohort study of IP-10's potential as a biomarker to aid in inflammation regulation within a clinical decision support protocol for patients with severe COVID-19. PLoS One. 2021 Jan 12;16(1):e0245296. doi: 10.1371/journal.pone.0245296. eCollection 2021. PMID 33434221